CLINICAL TRIAL: NCT05457582
Title: PCSK 9 Inhibitor Added to High-Intensity Statin Therapy to Prevent Cardiovascular Events in Patients With Acute Coronary Syndrome After Percutaneous Coronary Intervention: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study
Brief Title: PCSK 9 Inhibitor Added to High-Intensity Statin Therapy to Prevent Cardiovascular Events in Patients With ACS After PCI
Acronym: SHAWN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Collaborators: National Natural Science Foundation of China (Other Government); Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Shaoliang Chen, MD, Vice President of Nanjing First Hospital, Director of Cardiovascular Department, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NMU20220701
Record Dates: First submitted 2022-07-07; First posted 2022-07-14 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Acute Coronary Syndrome; Hyperlipidemias; Percutaneous Coronary Intervention; Cardiovascular Events
MeSH Terms: conditions — Acute Coronary Syndrome; Hyperlipidemias

STUDY DESIGN:
Intervention Model Description: Participants are randomly (at a ratio of 1:1) assigned to PCSK9 inhibitor plus high-intensity statin or placebo plus high-intensity statin group, and then the results at 1 year, 2- or 3-year are compared
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Neither the participants nor the investigators are aware of the treatment assignment until the end of the trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo plus high-intensity statin (Placebo Comparator): Participants received placebo subcutaneous injections once every 2 weeks (Q2W) plus high-intensity statin treatment (Rosuvastatin, 20 mg, once daily)
  Interventions: Drug: Placebo plus high-intensity statin
- PCSK 9 Inhibitor plus high-intensity statin (Active Comparator): Participants received PCSK 9 Inhibitor Q2W subcutaneous injections
  Interventions: Drug: PCSK 9 Inhibitor plus high-intensity statin

INTERVENTIONS:
Drug: Placebo plus high-intensity statin — Administered subcutaneously using a spring-based prefilled 1.0 mL autoinjector/pen, Q2W, and oral administration of rosuvastatin (20 mg, once daily).
  Arms: Placebo plus high-intensity statin
Drug: PCSK 9 Inhibitor plus high-intensity statin — Administered subcutaneously using a spring-based prefilled 1.0 mL autoinjector/pen, Q2W, and oral administration of rosuvastatin (20 mg, once daily).
  Arms: PCSK 9 Inhibitor plus high-intensity statin

SUMMARY:
The primary objective was to evaluate the effect of PCSK 9 Inhibitor (initiated within 4 h from PCI for the culprit lesion) with high-intensity statin treatment, compared to placebo with high-intensity statin treatment, on cardiovascular events (including cardiovascular death, myocardial infarction, stroke, re-hospitalization due to acute coronary syndromes or heart failure, or any ischemia-driven coronary revascularization) in patients with acute coronary syndrome and multiple lesions. Alirocumab was used before June 10, 2025; Tafolecimab has been used from June 10, 2025 onward.

DETAILED DESCRIPTION:
Patients with acute coronary syndrome (ACS) are at high-risk. ACS patients are commonly associated with multiple lesions or multivessel disease. Percutaneous coronary intervention (PCI) is an effective treatment for culprit lesions in ACS. Statin at high-intensity is recommended by current guidelines in order to prevent/slow the progression of non-culprit disease or restenosis. PCSK9 inhibitor serves as the most powerful medication in lowering LDL via promoting the expression of LDL receptors in the liver. However, if the combination of PCSK9 inhibitor with high-intensity statin treatment could significantly reduce the cardiovascular events in patients with ACS who underwent PCI remains unknown. Alirocumab was used before June 10, 2025; Tafolecimab has been used from June 10, 2025 onward.

ELIGIBILITY:
Inclusion Criteria:

1. The subject, or their legal guardian, must have a clear understanding of the trial's design and treatment procedures. They must provide written informed consent before any trial-specific tests or procedures are conducted.
2. Both male and female subjects aged ≥18 years.
3. Subjects who have experienced an ACS and have undergone PCI for culprit lesions (either QFR or FFR < 0.8) are eligible. ACS is defined as:

(1) Unstable angina (characterized by rest pain lasting between 5 and 30 minutes or worsening exertional angina accompanied by either transient ST segment depression or elevation, or angiography revealing visually estimated diameter stenosis of 90% or greater, or a ruptured plaque or thrombotic lesion), or (2) Non-ST elevation myocardial infarction, indicated by positive troponin levels consistent with the clinical syndrome and non-ST segment elevation, or (3) ST elevation myocardial infarction, indicated by positive troponin levels consistent with the clinical syndrome and ST-segment elevation.

4. Low-density lipoprotein cholesterol levels must meet the following criteria:

1. Low-density lipoprotein cholesterol ≥70 mg/dL (≥1.8 mmol/L) in patients who have been on a stable high-intensity statin regimen for at least 4 weeks before enrollment.
2. Low-density lipoprotein cholesterol ≥90 mg/dL (≥2.3 mmol/L) in patients who have been on a moderate or low-intensity statin regimen before enrollment.
3. Low-density lipoprotein cholesterol ≥125 mg/dL (≥3.2 mmol/L) in patients who are statin-naïve or have not been on a stable statin regimen for at least 4 weeks before enrollment.

5. Subjects must have at least one culprit lesion for ACS in a major native coronary artery (diameter stenosis >70% with a QFR or FFR<0.8), and have at least one non-culprit vessel disease (diameter stenosis ≤70% with a QFR or FFR ≥0.8).

Exclusion Criteria:

1. Fasting serum triglyceride levels exceeding 400 mg/dL (exceeding 4.52 mmol/L) before randomization.
2. Coronary artery disease is located within a saphenous vein graft or an arterial graft.
3. Residual diameter stenosis greater than 50% as determined by visual examination after percutaneous coronary intervention of the culprit lesion.
4. TIMI (Thrombolysis in Myocardial Infarction) flow less than 3 in the culprit vessel after PCI.
5. Unstable clinical status, characterized by hemodynamic (including cardiogenic shock) or electrical instability.
6. Uncontrolled hypertension, indicated by multiple readings with systolic blood pressure (SBP) exceeding 180 mmHg or diastolic blood pressure (DBP) exceeding 110 mmHg.
7. New York Heart Association (NYHA) Class III or IV, and an already known left ventricular ejection fraction (LVEF) below 30%.
8. Known history of hemorrhagic stroke in last 180 days before randomization.
9. Uncontrolled cardiac arrhythmia, defined as recurrent and symptomatic ventricular tachycardia or atrial fibrillation with rapid ventricular response that has not been controlled by medications in the past 3 months before screening.
10. Severe renal dysfunction, defined by an estimated glomerular filtration rate (eGFR) below 30 ml/min/1.73m².
11. Active liver disease or hepatic dysfunction.
12. Known intolerance to rosuvastatin or any statin.
13. Known allergy to contrast medium, heparin, aspirin, ticagrelor, prasugrel, or clopidogrel.
14. Subjects who have previously received PCSK9 inhibitors.
15. Subjects who have received cholesterol ester transfer protein inhibitors within the past 12 months before enrollment.
16. Treatment with systemic steroids or systemic cyclosporine within the past 3 months.
17. Known active infection or major hematologic, metabolic, or endocrine dysfunction, as determined by the Investigator.
18. Planned non-cardiac surgery within the next 12 months.
19. Subjects who will not be able to attend the required study visits, as determined by the Investigator.
20. Currently enrolled in another investigational device or drug study.
21. History of cancer within the past 5 years, unless adequately treated basal cell skin cancer, squamous cell skin cancer, or in situ cervical cancer.
22. Estimated life expectancy of less than 12 months.
23. Female of childbearing potential (age <50 years and last menstruation within the last 12 months), who did not undergo tubal ligation, ovariectomy, or hysterectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1212 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular events | 12 months after randomization
  Cardiovascular events defined as the composite of cardiovascular death, myocardial infarction, stroke or transit ischemic attack, re-hospitalization due to unstable angina or heart failure, or any ischemia-driven coronary revascularization.

SECONDARY OUTCOMES:
Cardiovascular death | 12 months after randomization
  It will be adjudicated by an independent external CEC according to protocol defined definition.
All cause death | 12 months after randomization
  It is defined as any death from randomization to the last visit.
Myocardial infarction | 12 months after randomization
  It will be adjudicated by an independent external CEC.
Stroke | 12 months after randomization
  stroke will be adjudicated by an independent external CEC.
Ischemia-driven coronary revascularization | 12 months after randomization
  It will be adjudicated by an independent external CEC.
Re-hospitalization due to unstable angina or heart failure | 12 months after randomization
  It will be adjudicated by an independent external CEC.
Diagnostic malignant tumor | 12 months after randomization
  It will be adjudicated by an independent external CEC.
PCSK9 inhibitors or statin intolerance | 12 months after randomization
  It will be adjudicated by an independent external CEC.

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Liang Chen, MD, PhD, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No